CLINICAL TRIAL: NCT03004482
Title: Noninvasive Monitoring and Diagnosis of Physiologic Disturbances in Term and Preterm Newborns Using Video Analysis Techniques
Brief Title: Analysis of Video Imaging in Newborns
Status: Suspended | Type: Observational
Why Stopped: lack of Funding
Sponsor: American University of Beirut Medical Center (Other)
Collaborators: Lebanese University (Other)
Responsible Party: Principal Investigator, Lama Charafeddine, Associate Professor of Clinical Pediatrics, American University of Beirut Medical Center
Other Study IDs: PED.LC.06
Record Dates: First submitted 2016-12-20; First posted 2016-12-29 (Estimated); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Neonatal Intensive Care Unit
Keywords: NICU; Recorded video images; physiological disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Video recording for term and preterm newborns hosted at the AUBMC Neonate ICU will be collected. The videos will capture movements, skin color changes, positioning, and other features relevant to the diagnosis in question. Recorded video images will be analysed by a computer software using the Eulerian Video magnification technology; then images will be correlated with simultaneously recorded physiological parameters (heart rate, respiratory rate and saturation). Images will be annotated by the clinician. Correlation between the skin coloration differentials and annotated physiological parameters may establish physiological indices. These may be used to extrapolate the existence or absence of disease states.

DETAILED DESCRIPTION:
Recent medical and technological advancements are progressively leading to increased survival rates of term and premature neonates. This project is concerned with detecting early signs of physiological disorders in term and preterm babies based on Eulerian Video Magnification, statistical analysis, and expert knowledge. Video recordings of skin coloration differentials for normal and sick neonates may be used to establish norms for each of the two major populations. Those and possibly other features will be used to develop an automatic contactless, noninvasive monitoring and diagnostic system that may detect early signs of disease. Early detection may lead to early diagnosis and preemptive treatment resulting in better outcome and lower costs of medical intervention. The objective of this project is to adapt the Eulerian Video Magnification for monitoring physiologic changes and then diagnosing potential disturbances in term and preterm neonates of different gestational ages. EVM uses video recordings of magnified skin color signals over time and thus permits analysis of physiological state changes such as heart rate and perfusion. Those changes would then be correlated with particular condition or disease states for the purpose of automatic early diagnosis and alarm issuance. Being contactless and non-invasive, the proposed system would be particularly helpful in vulnerable populations such as sick neonates. It may lead to earlier treatment, improved outcome, and possibly, decreased hospital stay.

Parents of infants admitted to the neonatal intensive care unit (NICU) at AUBMC will be informed about the study by their Attending physician. The medical research assistant will approach only interested and potential participants. An informed consent will be obtained prior to enrollment. All infants admitted to the NICU are eligible. Those will be divided into four equal groups: 1) "normal" term, 2) "normal" preterm, 3) "sick" term, and 4) "sick" preterm babies, where a "normal" health state is defined by the medical team as "physiologically stable". The medical team considers "sick" state based on pathological symptoms such as bradycardia, apnea, and hypotension among others. We target collecting video recordings for a total of eighty babies as a pilot number over the period of eight months. Each baby will be recorded for a minimum of twenty four hours. A subset of the eighty babies will be considered as a control group for reference. The control group will be selected based on a normal physiological state excluding babies with sepsis, respiratory distress, and congenital anomalies.

ELIGIBILITY:
Inclusion Criteria:

* Babies admitted to the neonatal intensive care unit (NICU) at AUBMC.

Exclusion Criteria:

* Babies with sepsis, respiratory distress, and congenital anomalies.

Ages: 1 Hour to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Term and preterm newborns hosted at the AUBMC Neonatal ICU.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2015-09; Primary Completion 2023-01 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Adaptation of the Eulerian Video Magnification monitoring technique for healthy term and preterm neonates. | 2 years
  Using EVM technology, variations in magnified skin color differentials will be used to establish norms by correlating image variation signals with physiological parameters in healthy infants.

SECONDARY OUTCOMES:
Adaptation of the Eulerian Video Magnification monitoring technique for diseased term and preterm neonates. | 2 years
  Using EVM technology, variations in magnified skin color differentials in diseased infants will be compared to the previously establish norms in order to permit early detection of changes in the physiological parameters in diseased infants.

CONTACTS AND LOCATIONS:
Overall Officials: Lama Charafeddine, MD FAAP, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aarts LA, Jeanne V, Cleary JP, Lieber C, Nelson JS, Bambang Oetomo S, Verkruysse W. Non-contact heart rate monitoring utilizing camera photoplethysmography in the neonatal intensive care unit - a pilot study. Early Hum Dev. 2013 Dec;89(12):943-8. doi: 10.1016/j.earlhumdev.2013.09.016. Epub 2013 Oct 14. PMID 24135159
- [Background] H.-Y. Wu, M. Rubinstein, E. Shih, J. Guttag, F. Durand, and W. T. Freeman. Eulerian video magnification for revealing subtle changes in the world. ACM Transactions on Graphics, 31(4), 2012.
- [Background] Edmond K, Zaidi A. New approaches to preventing, diagnosing, and treating neonatal sepsis. PLoS Med. 2010 Mar 9;7(3):e1000213. doi: 10.1371/journal.pmed.1000213. PMID 20231868
- [Background] Poh MZ, McDuff DJ, Picard RW. Non-contact, automated cardiac pulse measurements using video imaging and blind source separation. Opt Express. 2010 May 10;18(10):10762-74. doi: 10.1364/OE.18.010762. PMID 20588929
- [Background] Wynn JL, Wong HR. Pathophysiology and treatment of septic shock in neonates. Clin Perinatol. 2010 Jun;37(2):439-79. doi: 10.1016/j.clp.2010.04.002. PMID 20569817
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Background] Fairchild KD, Schelonka RL, Kaufman DA, Carlo WA, Kattwinkel J, Porcelli PJ, Navarrete CT, Bancalari E, Aschner JL, Walker MW, Perez JA, Palmer C, Lake DE, O'Shea TM, Moorman JR. Septicemia mortality reduction in neonates in a heart rate characteristics monitoring trial. Pediatr Res. 2013 Nov;74(5):570-5. doi: 10.1038/pr.2013.136. Epub 2013 Aug 13. PMID 23942558
- [Background] Moorman JR, Carlo WA, Kattwinkel J, Schelonka RL, Porcelli PJ, Navarrete CT, Bancalari E, Aschner JL, Whit Walker M, Perez JA, Palmer C, Stukenborg GJ, Lake DE, Michael O'Shea T. Mortality reduction by heart rate characteristic monitoring in very low birth weight neonates: a randomized trial. J Pediatr. 2011 Dec;159(6):900-6.e1. doi: 10.1016/j.jpeds.2011.06.044. Epub 2011 Aug 24. PMID 21864846
- [Background] Sullivan BA, Grice SM, Lake DE, Moorman JR, Fairchild KD. Infection and other clinical correlates of abnormal heart rate characteristics in preterm infants. J Pediatr. 2014 Apr;164(4):775-80. doi: 10.1016/j.jpeds.2013.11.038. Epub 2014 Jan 10. PMID 24412138
- [Background] K. J., B. S., G. G., and D. J. Non-contact heart rate and heart rate variability measurements. Biomedical signal processing and control, 13:102-112, 2014.
- [Background] Sztajzel J. Heart rate variability: a noninvasive electrocardiographic method to measure the autonomic nervous system. Swiss Med Wkly. 2004 Sep 4;134(35-36):514-22. doi: 10.4414/smw.2004.10321. PMID 15517504
- [Background] Kattwinkel J, Perlman JM, Aziz K, Colby C, Fairchild K, Gallagher J, Hazinski MF, Halamek LP, Kumar P, Little G, McGowan JE, Nightengale B, Ramirez MM, Ringer S, Simon WM, Weiner GM, Wyckoff M, Zaichkin J. Part 15: neonatal resuscitation: 2010 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2010 Nov 2;122(18 Suppl 3):S909-19. doi: 10.1161/CIRCULATIONAHA.110.971119. No abstract available. PMID 20956231
- [Background] Marodi L. Neonatal innate immunity to infectious agents. Infect Immun. 2006 Apr;74(4):1999-2006. doi: 10.1128/IAI.74.4.1999-2006.2006. No abstract available. PMID 16552028
- [Background] Liu L, Johnson HL, Cousens S, Perin J, Scott S, Lawn JE, Rudan I, Campbell H, Cibulskis R, Li M, Mathers C, Black RE; Child Health Epidemiology Reference Group of WHO and UNICEF. Global, regional, and national causes of child mortality: an updated systematic analysis for 2010 with time trends since 2000. Lancet. 2012 Jun 9;379(9832):2151-61. doi: 10.1016/S0140-6736(12)60560-1. Epub 2012 May 11. PMID 22579125
- [Background] Young Infants Clinical Signs Study Group. Clinical signs that predict severe illness in children under age 2 months: a multicentre study. Lancet. 2008 Jan 12;371(9607):135-42. doi: 10.1016/S0140-6736(08)60106-3. PMID 18191685
- [Background] Lozano R, Naghavi M, Foreman K, Lim S, Shibuya K, Aboyans V, Abraham J, Adair T, Aggarwal R, Ahn SY, Alvarado M, Anderson HR, Anderson LM, Andrews KG, Atkinson C, Baddour LM, Barker-Collo S, Bartels DH, Bell ML, Benjamin EJ, Bennett D, Bhalla K, Bikbov B, Bin Abdulhak A, Birbeck G, Blyth F, Bolliger I, Boufous S, Bucello C, Burch M, Burney P, Carapetis J, Chen H, Chou D, Chugh SS, Coffeng LE, Colan SD, Colquhoun S, Colson KE, Condon J, Connor MD, Cooper LT, Corriere M, Cortinovis M, de Vaccaro KC, Couser W, Cowie BC, Criqui MH, Cross M, Dabhadkar KC, Dahodwala N, De Leo D, Degenhardt L, Delossantos A, Denenberg J, Des Jarlais DC, Dharmaratne SD, Dorsey ER, Driscoll T, Duber H, Ebel B, Erwin PJ, Espindola P, Ezzati M, Feigin V, Flaxman AD, Forouzanfar MH, Fowkes FG, Franklin R, Fransen M, Freeman MK, Gabriel SE, Gakidou E, Gaspari F, Gillum RF, Gonzalez-Medina D, Halasa YA, Haring D, Harrison JE, Havmoeller R, Hay RJ, Hoen B, Hotez PJ, Hoy D, Jacobsen KH, James SL, Jasrasaria R, Jayaraman S, Johns N, Karthikeyan G, Kassebaum N, Keren A, Khoo JP, Knowlton LM, Kobusingye O, Koranteng A, Krishnamurthi R, Lipnick M, Lipshultz SE, Ohno SL, Mabweijano J, MacIntyre MF, Mallinger L, March L, Marks GB, Marks R, Matsumori A, Matzopoulos R, Mayosi BM, McAnulty JH, McDermott MM, McGrath J, Mensah GA, Merriman TR, Michaud C, Miller M, Miller TR, Mock C, Mocumbi AO, Mokdad AA, Moran A, Mulholland K, Nair MN, Naldi L, Narayan KM, Nasseri K, Norman P, O'Donnell M, Omer SB, Ortblad K, Osborne R, Ozgediz D, Pahari B, Pandian JD, Rivero AP, Padilla RP, Perez-Ruiz F, Perico N, Phillips D, Pierce K, Pope CA 3rd, Porrini E, Pourmalek F, Raju M, Ranganathan D, Rehm JT, Rein DB, Remuzzi G, Rivara FP, Roberts T, De Leon FR, Rosenfeld LC, Rushton L, Sacco RL, Salomon JA, Sampson U, Sanman E, Schwebel DC, Segui-Gomez M, Shepard DS, Singh D, Singleton J, Sliwa K, Smith E, Steer A, Taylor JA, Thomas B, Tleyjeh IM, Towbin JA, Truelsen T, Undurraga EA, Venketasubramanian N, Vijayakumar L, Vos T, Wagner GR, Wang M, Wang W, Watt K, Weinstock MA, Weintraub R, Wilkinson JD, Woolf AD, Wulf S, Yeh PH, Yip P, Zabetian A, Zheng ZJ, Lopez AD, Murray CJ, AlMazroa MA, Memish ZA. Global and regional mortality from 235 causes of death for 20 age groups in 1990 and 2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2095-128. doi: 10.1016/S0140-6736(12)61728-0. PMID 23245604